CLINICAL TRIAL: NCT06743997
Title: A Randomized, Open Label, Single Subcutaneous Dose, 2x2 Crossover Study to Investigate the Relative Bioavailability, Safety and Tolerability Among Different Eutropin Formulations in Healthy Volunteers
Brief Title: A Study to Compare Eutropin Formulations in Healthy Volunteers for Bioavailability, Safety, and Tolerability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LG-HGCL011
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Experimental): Participants receive a single subcutaneous dose of the Test Drug(T), in the first period, followed by a washout period, and then a single subcutaneous dose of the Reference Drug(R) in the second period.
  Interventions: Drug: Test Drug (Eutropin Catridge, 48IU/Cartridge); Drug: Reference Drug (Eutropin, 4 IU/vial)
- Sequence 2 (Experimental): Participants receive a single subcutaneous dose of the Reference Drug(R), in the first period, followed by a washout period, and then a single subcutaneous dose of the Test Drug(T) in the second period.
  Interventions: Drug: Test Drug (Eutropin Catridge, 48IU/Cartridge); Drug: Reference Drug (Eutropin, 4 IU/vial)

INTERVENTIONS:
Drug: Test Drug (Eutropin Catridge, 48IU/Cartridge) — Liqid somatropin
  Other Names: T; Test Drug
Drug: Reference Drug (Eutropin, 4 IU/vial) — Lyophilized somatropin
  Other Names: R; Reference Drug

SUMMARY:
A randomized, Open Label, Single Subcutaneous Dose, 2x2 Crossover Study to Investigate the Relative Bioavailability, Safety and Tolerability among Different Eutropin Formulations in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to 40years at screening.
* Voluntarily decide to participate and provide written informed consent.
* Able to receive the investigational product (IP) and pre-treatment drugs.
* Wiliing and able to comply with study requirements, including follow-up visits and blood/urine sampling.

Exclusion Criteria:

* History of conditions contraindicating somatropin or pre-treatment drugs.
* Clinically significant medical history.
* Participation in another clinical trial and receipt of an investigational product within 80 days prior to the first IP administration.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
AUClast of somatropin | 0 to 24 hours post-dose
  AUClast will be used to evaluate the pharmacokinetics of somatropin

SECONDARY OUTCOMES:
AUCinf of somatropin | 0 to 24 hours post-dose
  AUCinf will be used to evaluate the pharmacokinetics of somatropin.
Cmax of somatropin | 0 to 24 hours post-dose
  Cmax will be used to evaluate the pharmacokinetics of somatropin.
Tmax of soatropin | 0 to 24 hours post-dose
  Tmax will be used to evaluate the pharmacokinetics of somatropin.
T1/2β of somatropin | 0 to 24 hours post-dose
  T1/2β will be used to evaluate the pharmacokinetics of somatropin.
Change in IGF-1 levels | 0 to 24 hours post-dose
  Change in IGF-1 levels will be used to evaluate the parmacodynamic effect of somatropin.
Change in IGFBP-3 levels | 0 to 24 hours post-dose
  Change in IGFBP-3 levels will be used to evaluate the parmacodynamic effect of somatropin.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea